CLINICAL TRIAL: NCT00330694
Title: Efficiency of Physiotherapeutic Care in Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Dr M Munneke, UMC St Radboud, Neurology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 945-04-357
Record Dates: First submitted 2006-05-24; First posted 2006-05-29 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Parkinson's Disease
Keywords: Physical Therapy; Organisation of care
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Implementation of ParkNet within 8 regions
  Interventions: Other: ParkNet
- II (Other): Usual Care in 8 regions
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: ParkNet — Development of a network of dedicated physiotherapist with specific expertise in Parkinson's Disease and structured referrals to these ParkNet therapists by neurologists.
  Arms: I
Other: Usual Care — No altered organisation of physiotherapy care in Parkinson's Disease
  Arms: II

SUMMARY:
In the course of their disease, most patients with Parkinson's Disease (PD) face mounting mobility deficits, including difficulties with walking, balance, posture and transfers. This frequently leads to (fear of) falls, injuries, loss of independence, and inactivity which causes social isolation and increases the risk of osteoporosis or cardiovascular disease. These mobility deficits are difficult to treat with drugs and neurosurgery. However, physiotherapy is deemed effective in improving mobility deficits in PD. Physiotherapy is widely prescribed for this purpose in the Netherlands. Yet, the efficiency of current "usual care" physiotherapy can be questioned, for two reasons. First, the referral process seems inadequate because patients are mainly referred by neurologists who often lack insight into the (im-)possibilities of physiotherapy for PD. Consequently, patients with a real need for physiotherapy are not always referred (undertreatment), whereas others without a real need are (overtreatment). Furthermore, most therapists treating PD patients are not specifically trained in treating these patients. This is not surprising because average therapists rarely treat more than two patients per year in their practice. Therefore, patients who are being referred probably receive suboptimal treatment.

The objective of this study is to evaluate whether the efficiency of physiotherapeutic care for patients with Parkinson's disease can be improved, at a reduced cost, by targeting two key elements of the current care system: a) inadequate referral by neurologists; b) suboptimal treatment by physiotherapists. We expect that optimal referral combined with expert treatment will increase the efficiency, as reflected by increased health benefits for patients at equal or reduced costs'.

DETAILED DESCRIPTION:
Design In a Cluster Randomised Trial, 16 clusters will be randomly allocated to either network care (8 clusters with an altered organisation of physiotherapeutic care) or usual care (8 clusters with unchanged organisation of physiotherapeutic care). Clusters are formed by all PD patients living in the communities connected to participating regional hospitals in the 16 clusters.

The health care intervention in the experimental group has two elements: (a) an improved quality of referrals by neurologists; and (b) an improved quality of interventions by physiotherapists. Brief description Network Care: In each of the Network Care clusters, 5 to 7 motivated therapists are selected to enroll in a regional ParkNet and consequently trained. Training is focused at correct use of the evidence-based guidelines for physiotherapy in PD (Keus et al, 2006). This training consists of a 5-day competence-oriented course, web-based continues education supported by seminars, and use of a PD specific electronic patient record. Neurologists are informed about indications for referral to physiotherapy. Improved communication between neurologist and ParkNet therapists is initiated and supported.

Following implementation of the health care change, PD patients attending the neurological outpatient clinics of the individual hospitals within the clusters will be asked to participate. During a period of 6 months, PD patients will enrol in the study. Enrollees will be followed for 6 months to measure the use and quality of physiotherapy, patient health benefit and satisfaction, and costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic PD, diagnosed according to the Brain Bank criteria of the UK Parkinson's Disease Society
* Living independently in the community
* Able to complete the trial questionnaires.

Exclusion Criteria:

* Atypical parkinsonian syndromes
* Hoehn & Yahr stage 5
* Severe cognitive impairment
* Presence of major psychiatric disorders
* Severe co-morbidity (e.g. cancer) that interferes with daily functioning.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2006-05; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Modified MACTAR scale | 6 months

SECONDARY OUTCOMES:
Parkinson Activity Scale (secondary) | 6 months
Costs | 6 months
Proportion of correct referrals (tertiary) | 6 months
Quality of physiotherapy(tertiary) | 6 months
Incidence of Falls (tertiary) | 6 months
ALDS (tertiary) | 6 months
SF-36 (tertiary) | 6 months
EQ-5D (tertiary) | 6 months
Satisfaction of patients and professionals (tertiary) | 6 months
Self Assessment Disability Scale (tertiary) | 6 months
Freezing of Gait Questionnaire {tertiary} | 6 months
6 meter walk test {tertiary} | 6 months
4x3 meter walk test (tertiary) | 6 months
Single leg stance (tertiary) | 6 months
Posture and Gait score (tertiary) | 6 months
Timed Up and Go (tertiary) | 6 months
Falls Efficacy Scale {tertiary} | 6 months
9-hole pegboard test {tertiary} | 6 months
Health Anxiety and Depression Scale (tertiary) | 6 months
Physical activities assessed with the LAPAQ questionnaire (tertiary) | 6 months
Caregiver burden assessed with the Care Giver Strain Index (tertiary) | 6 months
PDQ-39 (Mobility Scale) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marten Munneke, PhD, Principal Investigator — UMC st Radboud; Bastiaan R Bloem, MD, PhD, Principal Investigator — UMC st Radboud
Locations (18):
- Netherlands (18):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Medisch Centrum Alkmaar, Alkmaar
  - Gelre Ziekenhuis, Apeldoorn
  - Ziekenhuis Gooi Noord, Blaricum
  - Reinier de Graaf Groep, Delft
  - Slingeland Ziekenhuis, Doetinchem
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - Groene Hart Ziekenhuis, Gouda
  - Kennemer Gasthuis, Haarlem
  - Ziekenhuis Hilversum, Hilversum
  - Westfries Gasthuis, Hoorn
  - Ziekenhuis Bernhoven, Oss
  - Medisch Centrum Haaglanden, Westeinde, The Hague
  - Viecurie Medisch Centrum, Venlo
  - 't Lange land ziekenhuis, Zoetermeer
  - Gelre Ziekenhuizen, Zutphen

REFERENCES:
- [Derived] Munneke M, Nijkrake MJ, Keus SH, Kwakkel G, Berendse HW, Roos RA, Borm GF, Adang EM, Overeem S, Bloem BR; ParkinsonNet Trial Study Group. Efficacy of community-based physiotherapy networks for patients with Parkinson's disease: a cluster-randomised trial. Lancet Neurol. 2010 Jan;9(1):46-54. doi: 10.1016/S1474-4422(09)70327-8. Epub 2009 Dec 1. PMID 19959398